CLINICAL TRIAL: NCT03824730
Title: Endovascular Treatment of Different Types of Aorto-iliac Occlusions
Brief Title: Endovascular Treatment of Aorto-iliac Occlusions
Status: Completed | Type: Observational
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Vladimir Cvetic, Principal Investigator, Clinical Centre of Serbia
Other Study IDs: CCSerbia Vasc
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Aorto-Iliac Occlusive Disease; Iliac Artery Occlusion; Iliac Artery Disease
Keywords: endovascular; stent; aorto-iliac; occlusions; iliac
MeSH Terms: conditions — Bites and Stings | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endovascular occlusions group: Group of patients with aorto-iliac occlusive disease (TASC B, C, D) in whom stenting of the Common and/or External Iliac Arteries were performed
  Interventions: Device: Stenting of the Common and/or External Iliac Arteries

INTERVENTIONS:
Device: Stenting of the Common and/or External Iliac Arteries — Stenting of the Common and/or External Iliac Arteries was performed in the angiographic suite. Under local anesthesia, arterial access was obtained through standard percutaneous puncture of the common femoral artery, brachial approach, or simultaneous brachial and femoral approach.
  Iliac lesion crossing was achieved through intraluminal or subintimal manner depending on the behavior of the lesion intraoperatively.
  Predilatation of the occlusion before stent deployment was performed at the discretion of the operator.
  Balloon-expandable stents were used for proximal, ostial lesions, whereas self-expanding stents were deployed in all other lesions.
  Both stents were used in long lesions involving heavily calcified common iliac arteries.
  Other Names: Percutaneous Transluminal Angioplasty; stent implantation

SUMMARY:
This study compares early and long-term results of the endovascular treatment among patients with different types of aorto-iliac occlusions.

DETAILED DESCRIPTION:
Endovascular treatment has been increasingly applied as a therapeutic option for aorto-iliac occlusive disease during the last decade, becoming the first-line treatment for many of the Trans-Atlantic Inter-Society Consensus document II (TASC II) categories. TASC II document in 2007 stated endovascular treatment as the method of choice up to type B occlusions and surgery for low-risk patients with type C and D occlusions, emphasizing that the patient's comorbidities as well as the operator's long-term success rates should be included in the decision-making process.

Revision of TASC II document in 2015 is suggesting that the preferred revascularization method should be based on each vascular center's competence and experience with the anatomic complexity, considering patient comorbidity and overall prognosis, supporting the endovascular-first approach in all 4 different kinds of lesions in highly experienced centers.

These changes over time are based on expert opinions derived from smaller studies from high volume centers, and that they reflect both the widespread gain of endovascular experience and technical developments over the last 2 decades, leading to a rising number of centers providing an endovascular-first approach even in complex TASC C and D occlusions.

Rationale for offering endovascular-first option to patient with complex lesion would be low risk of complication and long-term patency.

Our intention is to compare early and long-term results of the endovascular treatment among patients with different types of aorto-iliac occlusions in two Serbian vascular centres.

ELIGIBILITY:
Inclusion Criteria:

* Patient has aorto-iliac occlusions type B, C & D according to TASC-II classification
* Patient suffers from severe claudication (Rutherford 3) or critical limb ischemia (Rutherford 4 and 5)
* Patients fulfilling criteria for endovascular treatment of aorto-iliac occlusion according to criteria of the participating centres.

Exclusion Criteria:

* Patients with associated abdominal or iliac aneurysm, restenotic lesions, acute thrombi or dissections,
* Patients who experienced an initial technical failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with endovascular stent due to aorto-iliac occlusions
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Primary artery/stent patency rate | 60 Months
  Patients were assumed primary patent if the target vessel had continuous flow without revascularization, bypass, or amputation.

SECONDARY OUTCOMES:
Primary assisted artery/stent patency rate | 60 months
  Primary assisted patency is defined as continuous flow assisted with a revascularization when the target vessel has restenosed (>70%) at any time post-procedure.
Secondary patency artery/stent rate | 60 months
  Secondary patency is defined as reestablishment of flow to distal arteries after 100% occlusion has occurred at the target vessel at any time post-procedure
Clinical success | 60 months
  During the follow-up period, the improvement of Rutherford classification 1 grade or more than 1 grade.
Number of participants with periprocedural complications: hematoma, bleeding, pseudoaneurysm, renal failure, myocardial infarction, stroke, mortality, thrombosis of the treated segment | 1 month
  Identification of serious adverse events requiring correction of therapy or surgery. Will be used physiological parameter and questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Z Sagic, Prof, Principal Investigator — Institute for Cardiovascular Diseases Dedinje
Locations (2):
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Institute for Cardiovascular Diseases Dedinje, Belgrade

IPD SHARING:
Plan to Share IPD: No